CLINICAL TRIAL: NCT04544579
Title: Endovascular Graft Anchoring Different Regions of Ascending Aorta in the Treatment of Ascending Aortic Dissection: a Prospective， Controlled and Multicenter Study
Brief Title: Endovascular Graft Anchoring Different Regions of Ascending Aorta in the Treatment of Ascending Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Medical Association (Network)
Collaborators: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zaiping Jing, Professor, Chinese Medical Association
Other Study IDs: https://orcid.org/0000-0002-07
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Ascending Aortic Dissection
MeSH Terms: conditions — Dissection, Ascending Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ascending aortic dissection patients: Ascending aortic dissection patients
  Interventions: Device: Stent grafts anchored in different areas

INTERVENTIONS:
Device: Stent grafts anchored in different areas — Endovascular repair of ascending aortic dissection patients with stent grafts anchored in different areas

SUMMARY:
Aortic dissection is a deadly and dangerous disease. About 28% of patients with ascending aortic dissection can't tolerate open surgical trauma caused by thoracotomy and cardiopulmonary bypass, and the prognosis is poor. Minimally invasive endovascular treatment has been applied in the treatment of descending aortic dissection. However, due to the special anatomical structure and high speed /pressure blood flow, the treatment of ascending aorta dissection has become an international difficulty.

DETAILED DESCRIPTION:
This study was designed combination of retrospective and prospective methods, and focused on distal false lumen Aneurysmal Expansion of Aortic Dissection (DAEAD) . To formulate clinical data for the risk assessment of DAEAD, and best intracavitary treatment or long-term efficacy evaluation, we combined the results of genetic testing, evaluating the missense mutation, computer simulation of blood flow dynamics analysis, and clinical imaging analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aortic dissection diagnosed by CTA;
* With indications for endovascular treatment
* The luminal graft anchor is required to be located in the ascending aorta.

Exclusion Criteria:

* Import difficult, such as external iliac artery diameter is less than 6 mm bilateral iliac, artery stenosis distortions;
* Patients with severe comorbidities, such as severe myocardial insufficient blood supply, heart failure, arrhythmia, severe renal dysfunction, and severe blood coagulation dysfunction;
* Patients with malignant tumor, or other serious illness, life expectancy of less than 1 year；
* Puncture local infection and high fever;⑤ within 1 month of the large area;
* Contrast media in patients with cerebrovascular accident or digestive tract hemorrhage patients with allergies;
* Aortic ulcer or aortic wall hematoma and other atypical dissection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical trial included a prospective study of patients admitted to the hospital with aortic dissection between October 2020 and September 2023 who were treated with an endoluminal graft after exclusion of surgical contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
success of operation | before December 2022
  The operation was completed successfully without complications.

CONTACTS AND LOCATIONS:
Overall Officials: Zaiping Jing, Professor, Principal Investigator — Vascular surgery, Changhai Hospital

REFERENCES:
- [Derived] Pei Y, Zhu H, Xiao Y, Zhou J, Jing Z. The Mini-Cross Prefenestration for Endovascular Repair of Aortic Arch Pathologies. Front Cardiovasc Med. 2022 Jan 11;8:745871. doi: 10.3389/fcvm.2021.745871. eCollection 2021. PMID 35087876